CLINICAL TRIAL: NCT07309107
Title: Impact of Deep Learning-Based Noise Reduction Algorithm on Visual Analysis and Centiloid Quantification in Reduced-Dose and, or Time Acquisition Amyloid PET Imaging
Brief Title: Deep Learning on Amyloid Positons Emission Tomography
Acronym: DEEPAMY
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2025PI190
Record Dates: First submitted 2025-11-24; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reducing injected dose and/or acquisition time in amyloid PET imaging would improve comfort, radiation safety and cost-effectiveness in diagnosis and follow-up of patients. This study evaluates the impact of a deep learning-based noise reduction algorithm on visual analysis and Centiloid quantification when simulating reduced injected doses of [18F]flutemetamol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with objective cognitive impairment,
* Referred to our department for a cerebral [¹⁸F]flutemetamol positron emission tomography scan between January 1, 2023 and July 1, 2025,

Exclusion Criteria:

* Patient have objected to the use of their data.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with objective cognitive impairment, referred to our department for a cerebral [¹⁸F]flutemetamol positron emission tomography scan between January 1, 2023 and July 1, 2025, will be included
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of a deep-learning noise reduction algorithm on visual analysis and centiloid quantification when simulating reduced injected doses of 18F-flutemetamol. | Day one
  Visual analysis of the cerebral [¹⁸F]flutemetamol PET images will be performed by two nuclear medicine specialists in a blinded manner, with a third reader acting as an arbitrator in case of disagreement, according to routine diagnostic criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine VERGER, MD, PhD, Principal Investigator — CHRU of NANCY